CLINICAL TRIAL: NCT04821349
Title: Role of the Artificial Intelligence in Capsule Endoscopy for the Identification of Small Bowel Lesions in Patients With Small Intestinal Bleeding ArtIC Study: Artificial Intelligence Capsule Endoscopy Study
Brief Title: Role of AI in CE for the Identification of SB Lesions in Patients With Small Intestinal Bleeding.
Acronym: ArtIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Collaborators: Humanitas Hospital, Italy (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Skane University Hospital (Other); Hospital Clinic of Barcelona (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Endo-Kapszula Magánorvosi Centrum (Industry); Szeged University (Other); Saint Antoine University Hospital (Other); Hospital Avicenne (Other); South Tyneside and Sunderland NHS Foundation Trust (Other); Northwick Park Hospital (Other); Hospices Civils de Lyon (Other); Royal Free Hospital NHS Foundation Trust (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ArtiC STUDY-NP4350 v.05 140920
Record Dates: First submitted 2021-03-12; First posted 2021-03-29 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2022-11

CONDITIONS: Iron Deficiency Anemia; Obscure Gastrointestinal Bleeding
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Capsule Endoscopy

STUDY DESIGN:
Masking Description: Each center will receive from another center anonymized patient videos that have been uploaded on an encrypted USB key. Indeed, expert gastroenterologists from each center will proceed with AI-assisted video reading without knowing which center the video comes from nor the results of the normal reading. Reading conditions are the same as for standard reading.
  Results from both normal and AI-assisted reading will be compared. In the case of significant disagreement between the results from conventional capsule endoscopy reading and AI-assisted reading (e.g. missed lesions), a consensus review for each center will be done. Any lesion shall be considered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): Standard reading Group vs AI-assisted reading Group
  Interventions: Device: Capsule endoscopy

INTERVENTIONS:
Device: Capsule endoscopy — A consecutive series of patients recruited by 12 European centers based on the indication of OGIB will undergo capsule endoscopy examination.
  Capsule endoscopy will be performed in each site according to local rules and requirements, and the study protocol will concern only the post-procedure analysis on reading modalities for each patient.

SUMMARY:
Capsule Endoscopy (CE) is a safe, patient friendly and easy procedure performed for the evaluation of gastrointestinal tract unable to be explored via conventional endoscopy. The most common indication to perform SBCE is represented by Suspected Small Bowel Bleeding (SSBB). According to the widest meta-analysis available in literature, SBCE shows a diagnostic yield in SSBB of about 60%, and angiodysplasias are the most relevant findings, accounting for 50% of patients undergoing SBCE for SSBB. Accordingly, it represents the first line examination in SSBB investigation for determining the source of bleeding, if primary endoscopy results negative. Despite its high clinical feasibility, the evaluation of CE-video-captures is one of the main drawbacks since it is time consuming and requests the reader to concentrate to not miss any lesion. In order to reduce reading time, several software have been developed with the aim to cut similar images and select relevant images. For example, automated fast reading software have demonstrated to significantly reduce reading time without impacting the miss rate in pathological conditions affecting diffusely the mucosa (as IBD lesions do). Not the same assumption can be taken for isolated lesions since several studies reported an unacceptable miss rate for such a detection modality. New advancements such as artificial intelligence made their appearance in recent years. Deep convolutional neural networks (CNNs) have demonstrated to recognize specific images among a large variety up to exceed human performance in visual tasks. A Deep Learning model has been recently validated in the field of Small Bowel CE by Ding et al. According to their data collected on 5000 patients, the CNN-based auxiliary model identify abnormalities with 99.88% sensitivity in the per patient analysis and 99.90% sensitivity in the per-lesion analysis. With this perspective, it is believable that AI applied to SBCE can significantly shorten the reading time and support physicians to detect available lesions without losing significant lesions, further improving the diagnostic yield of the procedure.

DETAILED DESCRIPTION:
This is a multicenter, multinational, blinded prospective trial, involving a consecutive series of patients recruited by 12 European centers based on the indication of OGIB:

* after negative upper and lower endoscopy
* France: after negative pregnancy test
* Hb cut-off male: <13, female: <12 Capsule endoscopy will be performed in each site according to local rules and requirements, and the study protocol will concern only the post-procedure analysis on reading modalities for each patient, as specified below.1. Regimen of preparation AI depends on the possibility of the software to "see" images. An inadequate cleansing level precludes a proper visualization and the impact of technology. In order to have homogenous results, a standard regimen of preparation is advisable. The regimen includes a split dose of PEG-based solution (PlenVu, Moviprep) as recommended by ESGE guideline - technical report. Dose 1 will be administered at 7 pm of the day before and dose 2 in the morning of the procedure in order to be completed at least 1 hour before capsule ingestion. On the day before patients can have breakfast and a light meal. After lunch they should be fasting. Two and 4 hours after capsule ingestion patient are allowed to drink clear liquids and a light meal, respectively.

  2. Standard reading Each center will review the images collected according to the "normal reading" as recommended by ESGE guidelines. To compare reading time correctly, readers must read the video without including annotation of images. All lesions should be considered independently of their relevance. Findings are not marked on every image if they appear repeatedly on every consecutive image, but if they appear repeatedly with normal images in between. Annotations should be done after the reading, each lesion shall be labelled if it belongs to P1/2 category according to the Saurin Classification. Definition of P1, P2: red spots on the intestinal mucosa or small or isolated erosions or angioectasia, ulcers, tumors or varices or any other bleeding abnormality.

  3. AI-assisted reading Each center will receive from another center anonymized patient videos that have been uploaded on an encrypted USB key. Indeed, expert gastroenterologists from each center will proceed with AI-assisted video reading without knowing which center the video comes from nor the results of the normal reading. Reading conditions are the same as for standard reading.

  4. Consensus reading Results from both normal and AI-assisted reading will be compared. In the case of significant disagreement between the results from conventional capsule endoscopy reading and AI-assisted reading (e.g. missed lesions), a consensus review for each center will be done. Any lesion shall be considered.

ELIGIBILITY:
Inclusion Criteria:

indication of OGIB:1)after negative upper and lower endoscopy; 2)France: after negative pregnancy test; 3)Hb cut-off male: <13, female: <12

Exclusion Criteria:

* Age < 18 years old
* Known or suspected intestinal obstruction
* Non-steroidal anti-inflammatory drugs (twice weekly or more) during the 4 weeks preceding enrollment
* Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule
* Patient with known gastrointestinal motility disorders
* Subjects with known or suspected delayed gastric emptying
* Patient suffers from any condition, such as swallowing problems, which precludes compliance with study and/or device instructions
* Patient has any allergy or other known contraindication or intolerance to the medications used in the study
* Patient has any condition, which precludes compliance with study and/or device instructions
* Patient with any contraindication to take the bowel preparation product
* Women who are either pregnant or nursing at the time of screening, or are of child- bearing potential and do not practice medically acceptable methods of contraception
* Concurrent participation in another clinical trial using any investigational drug or device
* Patient suffers from a life-threatening condition
* Patients with history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters
* Patients with pace-maker or implantable cardioverter
* Patient did not sign informed consent
* Endoscopic placement of the capsule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of AI-assisted video reading versus traditional video reading with conventional software. | through study completion, an average of 1 year
  sensitivity, specificity, PPV, NPV calculated at per-patient analysis for P1 / P2 lesions, compared with the adjudication committee as gold standard in case of discrepancies.

SECONDARY OUTCOMES:
evaluation of Reading time of AI-assisted reading compared with conventional reading | through study completion, an average of 1 year
Role of AI-assisted reading in real life from a health economic perspective | through study completion, an average of 1 year
Accuracy of AI-assisted video reading versus traditional video reading with conventional software. | through study completion, an average of 1 year
  Sensitivity, specificity, PPV, NPV, calculated at per lesion analysis for P1 / P2 lesions and for any lesion with the adjudication committee as gold standard in case of discrepancies .
Accuracy of AI-assisted video reading versus traditional video reading with conventional software considering any lesions for a per-patient analysis with the adjudication committee as gold standard in case of discrepancies. | through study completion, an average of 1 year
Diagnostic yield of CE | through study completion, an average of 1 year
Number and type of findings / lesion detected | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Poliambulanza, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
All data and source code can be made available after the manuscript publication on reasonable request, which must include an appropriate protocol, analysis plan, and data exchange with institutional approvals in place before data transfer of any information.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Spada C, Piccirelli S, Hassan C, Ferrari C, Toth E, Gonzalez-Suarez B, Keuchel M, McAlindon M, Finta A, Rosztoczy A, Dray X, Salvi D, Riccioni ME, Benamouzig R, Chattree A, Humphries A, Saurin JC, Despott EJ, Murino A, Johansson GW, Giordano A, Baltes P, Sidhu R, Szalai M, Helle K, Nemeth A, Nowak T, Lin R, Costamagna G. AI-assisted capsule endoscopy reading in suspected small bowel bleeding: a multicentre prospective study. Lancet Digit Health. 2024 May;6(5):e345-e353. doi: 10.1016/S2589-7500(24)00048-7. PMID 38670743